CLINICAL TRIAL: NCT00001782
Title: Hemispheric Lateralization of Language Receptive Function in the Deaf and in Hearing Individuals Who Learned ASL as First Language
Brief Title: Areas of Brain Responsible for Understanding American Sign Language
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980082; 98-N-0082
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-11

CONDITIONS: Brain Mapping; Deafness; Healthy
Keywords: Deafness; Hemisphere Dominance; Language; Plasticity; Speech; rTMS
MeSH Terms: conditions — Deafness; Language; Speech

SUMMARY:
The human brain is made up of two halves called hemispheres. Each half of the brain is responsible for processing different kinds of information. Previous neuroimaging studies have shown that both the right and left hemispheres are involved when processing information given in American Sign Language (ASL). However, the study also showed that when processing spoken language, the left hemisphere was mostly involved.

Researchers would like to find out more about how the brain processes American Sign Language (ASL). This study is designed to determine if the right hemisphere is necessary for normal understanding of ASL.

DETAILED DESCRIPTION:
The purpose of this protocol is to determine if the right hemisphere activation associated with perception of American Sign Language (ASL) in deaf subjects and in normal hearing individuals raised by deaf parents (who learned ASL before written English) is necessary for appropriate understanding of ASL.

ELIGIBILITY:
Subject age between 18 and 65 years.

Adult hearing offsprings of deaf parents.

Congenitally deaf individuals.

Intact hearing volunteers.

No subjects with personal or family history of seizures or other neurological or demyelinating disorders.

No pregnant women tested after urine pregnancy test.

No subjects with severe coronary disease.

No subjects with metal in the cranium except mouth.

No subjects with intracardiac lines and implanted medication pumps.

No subjects with increased intracranial pressure as evaluated by clinical means.

No subjects with cardiac pacemakers.

No subjects with an intake of neuroleptics.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 1998-03; Study Completion 2000-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Neville HJ, Bavelier D, Corina D, Rauschecker J, Karni A, Lalwani A, Braun A, Clark V, Jezzard P, Turner R. Cerebral organization for language in deaf and hearing subjects: biological constraints and effects of experience. Proc Natl Acad Sci U S A. 1998 Feb 3;95(3):922-9. doi: 10.1073/pnas.95.3.922. PMID 9448260
- [Background] Cohen LG, Bandinelli S, Sato S, Kufta C, Hallett M. Attenuation in detection of somatosensory stimuli by transcranial magnetic stimulation. Electroencephalogr Clin Neurophysiol. 1991 Oct;81(5):366-76. doi: 10.1016/0168-5597(91)90026-t. PMID 1718723